CLINICAL TRIAL: NCT07211230
Title: Collagenase Producing Bacteria as a Biomarker and Driver of Diet-induce Colorectal Cancer Recurrence and Metastasis Following Surgery
Brief Title: Collagenase Biobank Study
Status: Not yet recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: University of California, San Diego (Other); Midwestern University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB25-0833
Record Dates: First submitted 2025-09-05; First posted 2025-10-07 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-06

CONDITIONS: Colorectal (Colon or Rectal) Cancer
Keywords: colorectal cancers; biobank; Collagenase Biobank; Tissue collection; stool collection
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected prior to surgery, day of surgery, during hospitalization, 6 months after surgery, and 12 months after surgery. The prior to surgery sample, during surgery, and during hospitalization samples will be collected as part of routine lab draws.
  Tissue Collection: A surgically resected malignant tumor tissue and adjacent normal tissue sample will be processed and created into organoids by the UChicago Organoid and Primary Culture Research Core (OPCR).
  Stool collection: For the preoperative and postoperative samples stool will be self-collected with a specimen kit that is provided to each patient at study enrollment. The patient will use this kit to collect and send stool specimens overnight at 4 degrees Celsius to PI Shogan's laboratory. For the inpatient sample, the sample will be collected by the nurse and a member of the research team will bring to the Shogan Lab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to look at how bacteria present within the stool at the time of surgery and postoperatively may contribute to the development of cancer recurrence after surgery. By collecting stool and blood before and after surgery, the researchers hope to determine if certain types of bacteria, or products that the bacteria produce, promote the development of tumors after surgery. By collecting tumor tissue and growing cell lines, we hope this will help researchers better understand the behavior of these types of tumors.

DETAILED DESCRIPTION:
The purpose of this study is to collect stool, blood, and tissue samples both before and after patients undergo surgery for colon cancer. These samples will be analyzed for their bacterial composition and function, and assayed for bacterial-derived metabolites. Additionally, these samples will be tested in the laboratory for their ability to promote tumor formation in cancer cells and in animal models of surgery. Finally, patients will undergo nutritional surveys to document their current nutritional intake. Integration of the patient's nutritional intake with the data from the analyzed biospecimens will allow the researchers to determine if these bacteria and/or their metabolites are more prevalent in patients who eat certain diets. Taken together, results from this study will provide knowledge as to the mechanisms by which tumors form after surgery and potentially allow for future therapies to prevent it.

ELIGIBILITY:
Inclusion Criteria:

* English speaking.
* All genders, races, and ethnicities.
* Aged greater or equal to 18 years of age.
* Ability to understand and the willingness to sign a written informed consent form.
* Diagnosed with a colon adenocarcinoma or presumed adenocarcinoma in which surgical resection is recommended.
* Have a planned surgical resection of the colon adenocarcinoma at the University of Chicago Comprehensive Cancer Center.
* Reside within 150 miles of the University of Chicago Comprehensive Cancer Center.

Exclusion Criteria:

* Stage IV colon adenocarcinoma (known metastatic disease).
* Intravenous or oral antibiotic exposure within 30 days of surgery to treat an infection.
* Prebiotic exposure within 30 days of surgery.
* History of neoadjuvant chemotherapy/radiation to treat the primary colon adenocarcinoma.
* History of chemotherapy/radiation to treat a separate malignancy within the last 6 months.
* History or current ileostomy or colostomy.
* Allergy to perioperative medications (oral neomycin/metronidazole for preoperative bowel preparation, intraoperative prophylactic intravenous cefoxitin).
* Patients who are pregnant.
* Patients with a history of inflammatory bowel disease.
* Patients with a history of bariatric surgery.
* History of eating disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing Colorectal Surgery
Sampling Method: Non-Probability Sample
Enrollment: 107 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Collagenase Activity | From Enrollment to 12 months postoperative.
  Measure collagenase activity present within the stool at the time of surgery to determine if it will be significantly higher in patients who later develop recurrence compared to patients who do not. Assessing further if patients who are the most nutritionally at risk for the development of recurrence will have the highest amounts of bacterial collagenase.

SECONDARY OUTCOMES:
Stool Metagenomics | From Enrollment to 12 months postoperative.
  Assess the correlation of the bacterial community with nutritional intake and the development of colorectal cancer recurrence. Bacterial community analysis will be performed via shotgun metagenomics.
Stool metabolomics | From Enrollment to 12 months postoperative.
  Assess the correlation of the bacterial derived metabolites with nutritional intake and the development of colorectal cancer recurrence. Bacterial community analysis will be performed via short chain fatty acid metabolomics.
Serum Metabolomics | From Enrollment to 12 months postoperative
  Assess the correlation of the bacterial derived metabolites with nutritional intake and the development of colorectal cancer recurrence. Bacterial community analysis will be performed via short chain fatty acid metabolomics.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin P Shogan, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States